CLINICAL TRIAL: NCT00438932
Title: Reduced Phosphate Intake in "Normo-Phosphatemic" Chronic Kidney Disease Patients
Brief Title: Low Phosphate Diets in Patients With Early Stages of Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Myles S. Wolf, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2005P000486
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Kidney Disease
Keywords: phosphate, phosphorus, FGF-23, PTH, 1,25D
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — lanthanum carbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lanthanum Carbonate and Low Phosphorus Diet (Active Comparator): 25% of subjects will receive binders plus a phosphate restricted diet.
  Interventions: Drug: Lanthanum Carbonate; Dietary Supplement: Low Phosphorus Diet
- Lanthanum Carbonate and Unrestricted Phosphorus Diet (Active Comparator): 25% binders + unrestricted phosphate diet.
  Interventions: Drug: Lanthanum Carbonate; Dietary Supplement: Unrestricted Phosphorus Diet
- Placebo and Low Phosphorus Diet (Active Comparator): 25% placebo + phosphate restricted diet.
  Interventions: Dietary Supplement: Low Phosphorus Diet; Drug: Placebo
- Placebo and Unrestricted Phosphorus Diet (Active Comparator): 25% placebo + unrestricted phosphate diet.
  Interventions: Dietary Supplement: Unrestricted Phosphorus Diet; Drug: Placebo

INTERVENTIONS:
Drug: Lanthanum Carbonate — Lanthanum carbonate 1000mg 3x/day
  Arms: Lanthanum Carbonate and Low Phosphorus Diet; Lanthanum Carbonate and Unrestricted Phosphorus Diet
Dietary Supplement: Low Phosphorus Diet — Low phosphorus diet will consist of 800 mg of phosphorus per day.
  Arms: Lanthanum Carbonate and Low Phosphorus Diet; Placebo and Low Phosphorus Diet
Dietary Supplement: Unrestricted Phosphorus Diet — Unrestricted diet will contain 1550 mg of phosphorus per day - 800 mg of which is dietary and 750mg of Neutraphos (3 packets/day); each packet is 250mg.
  Other Names: Neutraphos
  Arms: Lanthanum Carbonate and Unrestricted Phosphorus Diet; Placebo and Unrestricted Phosphorus Diet
Drug: Placebo — Lanthanum Carbonate placebo given three times a day with meals.
  Arms: Placebo and Low Phosphorus Diet; Placebo and Unrestricted Phosphorus Diet

SUMMARY:
The purpose of this study is to learn more about how the kidneys control the blood levels of phosphorus in patients with early chronic kidney disease. The ultimate goal is to use this information to design improved treatment strategies for phosphorus-related problems for the millions of patients with chronic kidney disease.

DETAILED DESCRIPTION:
Phosphorus is a mineral found in dairy products, nuts, and meat that is essential for bone health and many other important functions inside the body's cells. The kidneys are responsible for keeping the blood levels of phosphorus normal. Healthy kidneys do this by spilling excess phosphorus into the urine. In patients with chronic kidney disease, the kidneys are unable to spill an adequate amount of phosphorus so that excess phosphorus can accumulate in the walls of blood vessels leading to heart disease, their leading cause of death. A recently discovered hormone called FGF-23 helps control the blood levels of phosphorus by "telling" the kidney how much phosphorus to spill in the urine. The purpose of this study is to learn more about how FGF-23 helps the kidneys control the blood levels of phosphorus. The ultimate goal is to use this information to design improved treatment strategies for phosphorus-related problems for the millions of patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* subjects with stage 3a, 3b and 4 CKD
* subjects have to be aged 18 years or older
* subjects have to have normal serum phosphate levels (< 4.6 mg/dl)
* subjects have to have sufficient 25-OH Vit0amin D levels (≥ 20 ng/ml)

Exclusion Criteria:

* subjects with rapidly advancing renal failure who thus might develop hyperphosphatemia or end stage renal disease requiring initiation of dialysis during the study period
* subjects expected to require dialysis initiation within the follow up period
* subjects with hyperphosphatemia > 4.6 mg/dL
* subjects with any previous or current treatment with phosphate binders or active vitamin D (doxercalciferol or calcitriol)
* subjects with malnutrition, defined as a serum albumin < 3.0 mg/dl, in order to avoid worsening protein-malnutrition status during the restricted study period since phosphate restricted diets are also low in protein
* subjects with chronic gastrointestinal diseases that could impede their absorptive ability such as Crohn's disease, ulcerative colitis and sprue
* subjects with liver disease (ALT or AST > 100 U/L) or cholestasis (direct bilirubin > 1.0 mg/dl) because this can limit their ability to absorb fat soluble vitamins such as vitamin D
* subjects with anemia, defined as a hematocrit <27% at the screening visit
* subjects wht have been hospitalization within the previous 4 weeks
* subjects who are pregnant
* subjects who are breastfeeding mothers
* subjects with primary hypoparathyroidism
* subjects with primary hyperparathyroidism
* subjects with previous subtotal parathyroidectomy
* subjects with previous outpatient counseling by a renal nutritionist
* subjects who are unable to independently provide written informed consent - prisoners, mentally incompetent, minors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myles Wolf, MD, MMSc, Principal Investigator — Univesity of Miami Miller School of Medicine; Harald Jueppner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Isakova T, Gutierrez OM, Smith K, Epstein M, Keating LK, Juppner H, Wolf M. Pilot study of dietary phosphorus restriction and phosphorus binders to target fibroblast growth factor 23 in patients with chronic kidney disease. Nephrol Dial Transplant. 2011 Feb;26(2):584-91. doi: 10.1093/ndt/gfq419. Epub 2010 Jul 14. PMID 20631407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 patients completed the full study. Patients were recruited from renal clinics.
Pre-assignment Details: There was no wash-out, run in or transition.
Groups:
- Lanthanum Carbonate & Low Phosphorous Diet: Lanthanum carbonate 1000mg 3x/day and low phosphorus diet of 800 mg of phosphorus per day.
- Lanthanum Carbonate & Unrestricted Phosphorous Diet: Lanthanum carbonate 1000mg 3x/day and unrestricted diet containing 1550 mg of phosphorus per day - 800 mg of which is dietary and 750mg of Neutraphos (3 packets/day); each packet is 250mg.
- Placebo & Low Phosphorous Diet: Placebo and low phosphorus diet consisting of 800 mg of phosphorus per day.
- Placebo & Unrestricted Phosphorous Diet: Placebo and unrestricted diet containing 1550 mg of phosphorus per day - 800 mg of which is dietary and 750mg of Neutraphos (3 packets/day); each packet is 250mg.
Period: Overall Study
Arm/Group | Lanthanum Carbonate & Low Phosphorous Diet | Lanthanum Carbonate & Unrestricted Phosphorous Diet | Placebo & Low Phosphorous Diet | Placebo & Unrestricted Phosphorous Diet
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanthanum Carbonate & Low Phosphorous Diet | Lanthanum Carbonate & Unrestricted Phosphorous Diet | Placebo & Low Phosphorous Diet | Placebo & Unrestricted Phosphorous Diet | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 2 | 10
  >=65 years | 1 | 1 | 2 | 2 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (11) | 62 (13) | 56 (21) | 68 (17) | 62 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 1
  Male | 3 | 4 | 4 | 4 | 15
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 16
Fibroblast Growth Factor 23 (FGF-23) [Mean (Standard Deviation); unit: Ru/ml] — Plasma FGF-23 at the baseline visit was measured using C-terminal FGF23 assay.
  Ru/ml | 164.3 (110.9) [77 to 252] | 263.1 (167.9) [158 to 368] | 178.8 (97.6) [103 to 254] | 121.8 (60.0) [85 to 158] | 182.0 (116.3) [95 to 223]
24-hr urine phosphate [Mean (Standard Deviation); unit: mg] — measured from 24 hour urine collections; 2 separate collections were obtained; values are means of the two collections; pre-intervention
  mg | 659.0 (269.8) [491 to 827] | 761.8 (77.4) [704 to 820] | 745.4 (287.0) [503 to 988] | 934.6 (545.5) [607 to 1262] | 775.2 (320.0) [564 to 889]

OUTCOME MEASURES:

1. Primary Outcome: Fibroblast Growth Factor 23 (FGF-23)
Description: Plasma FGF-23 was measured using c-terminal FGF23 assay.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: RU/ml
Arm/Group | Lanthanum Carbonate & Low Phosphorous Diet | Lanthanum Carbonate & Unrestricted Phosphorous Diet | Placebo & Low Phosphorous Diet | Placebo & Unrestricted Phosphorous Diet
Number analyzed (Participants) | 4 | 4 | 4 | 4
RU/ml | 162.695 (56.170737) | 297 (77.69778) | 188.975 (60.2020815) | 143.7675 (37.507486)

2. Secondary Outcome: 24-hour Urinary Phosphate
Description: from 24-hr urine collections
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: mg
Arm/Group | Lanthanum Carbonate & Low Phosphorous Diet | Lanthanum Carbonate & Unrestricted Phosphorous Diet | Placebo & Low Phosphorous Diet | Placebo & Unrestricted Phosphorous Diet
Number analyzed (Participants) | 4 | 4 | 4 | 4
mg | 150.4 (49.3063045) | 382.725 (7.0577825) | 346.8 (132.671329) | 830.25 (220.003449)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Lanthanum Carbonate & Low Phosphorous Diet | Lanthanum Carbonate & Unrestricted Phosphorous Diet | Placebo & Low Phosphorous Diet | Placebo & Unrestricted Phosphorous Diet
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
In addition to limited power, the small sample size led to imbalances in baseline laboratory tests, which added further variability to the analyses. .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No